CLINICAL TRIAL: NCT00391443
Title: Effects of Bosentan on Morbidity and Mortality in Patients With Idiopathic Pulmonary Fibrosis - a Multicenter, Double-blind, Randomized, Placebo-controlled, Parallel Group, Event-driven, Group Sequential, Phase III Study.
Brief Title: BUILD 3: Bosentan Use in Interstitial Lung Disease
Acronym: BUILD 3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC-052-321
Record Dates: First submitted 2006-10-20; First posted 2006-10-24 (Estimated); Results first posted 2012-05-25 (Estimated); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: BUILD 3; Idiopathic Pulmonary Fibrosis; Tracleer; Interstitial Lung Disease; bosentan; Actelion
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Lung Diseases, Interstitial | interventions — Bosentan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Bosentan (Experimental): Subjects receive bosentan 62.5 mg twice daily (b.i.d.) for 4 weeks followed by bosentan 125 mg b.i.d (if body weight > 40 kg) or bosentan 62.5 mg b.i.d. (if body weight < 40 kg)
  Interventions: Drug: Bosentan
- Placebo (Placebo Comparator): Subjects receive placebo matching the bosentan treatment regimen
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bosentan — Bosentan 62.5 mg tablets twice daily (b.i.d.) for 4 weeks followed by bosentan 125 mg tablets b.i.d (if body weight > 40 kg) or bosentan 62.5 mg tablets b.i.d. (if body weight < 40 kg)
  Other Names: Ro 47-0203; ACT-050088
  Arms: Bosentan
Drug: Placebo — Placebo matching bosentan 62.5 mg tablets and 125 mg tablets
  Arms: Placebo

SUMMARY:
BUILD 3 is a prospective, multicenter, randomized, double-blind, parallel group, placebo-controlled, event-driven, group sequential, phase III superiority study. The primary objective is to demonstrate that bosentan delays disease worsening or death in patients with Idiopathic Pulmonary Fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Male or female aged 18 years or older (females of child-bearing potential must have been surgically sterilized or use a reliable method of contraception.)
* Proven diagnosis of IPF according to American Thoracic Society / European Respiratory Society (ATS-ERS) statement, of <3 years, with surgical lung biopsy (SLB)

Exclusion Criteria:

* Interstitial lung disease due to conditions other than IPF.
* Presence of extensive honeycombing (HC) on baseline high-resolution computed tomography (HRCT) scan.
* Severe concomitant illness limiting life expectancy (<1 year).
* Severe restrictive lung disease.
* Obstructive lung disease.
* Diffusing capacity of the lung for carbon monoxide <30% predicted.
* Residual volume > or = 120% predicted.
* Documented sustained improvement of patient's IPF condition up to 12 months prior to randomization with or without IPF-specific therapy.
* Recent pulmonary or upper respiratory tract infection (up to 4 weeks prior to randomization).
* Acute or chronic impairment (other than dyspnea) limiting the ability to comply with study requirements.
* Chronic heart failure with New York Heart Association (NYHA) class III/IV or known left ventricular ejection fraction <25%.
* Alanine aminotransferase (ALT/SGPT) and/or aspartate aminotransferase (AST/SGOT) > 1.5 times the upper limit of the normal ranges.
* Moderate to severe hepatic impairment.
* Serum creatinine > or = 2.5 mg/dl or chronic dialysis.
* Hemoglobin concentration <75% the lower limit of the normal ranges.
* Systolic blood pressure <85 mmHg.
* Pregnancy or breast-feeding.
* Current drug or alcohol dependence.
* Chronic treatment with the following drugs prescribed for IPF (within 4 weeks of randomization):oral corticosteroids (>20 mg/day of prednisone or equivalent), immunosuppressive or cytotoxic drugs, antifibrotic drugs, chronic use of N-acetylcysteine (prescribed for IPF).
* Oral anticoagulants other than those indicated for a venous or arterial thrombotic disease.
* Treatment with glibenclamide (glyburide) and calcineurin inhibitors (cyclosporine A, tacrolimus) up to 1 week prior to randomization.
* Treatment with an endothelin receptor antagonist up to 3 months prior to randomization.
* Participation in the BUILD 1 trial.
* Treatment with another investigational drug up to 3 months prior to randomization or planned treatment.
* Known hypersensitivity to bosentan or any of the excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 616 (Actual)
Dates: Start 2007-02; Primary Completion 2010-02 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Leconte, Study Director — Actelion

REFERENCES:
- [Derived] King TE Jr, Brown KK, Raghu G, du Bois RM, Lynch DA, Martinez F, Valeyre D, Leconte I, Morganti A, Roux S, Behr J. BUILD-3: a randomized, controlled trial of bosentan in idiopathic pulmonary fibrosis. Am J Respir Crit Care Med. 2011 Jul 1;184(1):92-9. doi: 10.1164/rccm.201011-1874OC. Epub 2011 Apr 7. PMID 21474646

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo; Bosentan: Initial dose: 62.5 mg twice daily (b.i.d.) for 4 weeks. Target dose: - body weight > 40 kg (90 lb): 125 mg b.i.d., (if the initial dose is well tolerated); - body weight < 40 kg (90 lb): 62.5 mg b.i.d.
Period: Overall Study
Arm/Group | Placebo | Bosentan
Started | 209 (1 patient in the bosentan arm did not receive treatment & was excluded from the Safety Population.) | 407
Completed | 209 | 407
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Bosentan | Total
Number analyzed (Participants) | 209 | 407 | 616
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (9.1) | 63.8 (8.4) | 63.6 (8.6)
Age, Customized [Number; unit: participants]
  Between 18 and 40 years | 4 | 5 | 9
  Between 41 and 60 years | 74 | 119 | 193
  Between 61 and 70 years | 87 | 195 | 282
  > 70 years | 44 | 88 | 132
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 111 | 187
  Male | 133 | 296 | 429
Region of Enrollment [Number; unit: participants]
  United States | 99 | 185 | 284
  Serbia | 2 | 0 | 2
  Spain | 7 | 15 | 22
  Ireland | 2 | 2 | 4
  Austria | 3 | 4 | 7
  Israel | 7 | 16 | 23
  Switzerland | 5 | 8 | 13
  Italy | 8 | 14 | 22
  United Kingdom | 3 | 7 | 10
  France | 9 | 14 | 23
  Czech Republic | 5 | 9 | 14
  Canada | 14 | 30 | 44
  Belgium | 1 | 2 | 3
  Croatia | 0 | 2 | 2
  Australia | 11 | 22 | 33
  Germany | 10 | 26 | 36
  Netherlands | 0 | 2 | 2
  Japan | 14 | 26 | 40
  Korea, Republic of | 9 | 23 | 32

OUTCOME MEASURES:

1. Primary Outcome: Time to Occurrence of Disease Worsening or Death up to End of Study.
Description: Disease worsening was defined as an event of worsening of pulmonary function tests (PFT) or acute exacerbation of idiopathic pulmonary fibrosis (IPF).
Time Frame: 36 months
Population: The primary analysis was performed on the Intent To Treat (ITT) population.
Measure: Number; unit: participants with event
Arm/Group | Placebo | Bosentan
Number analyzed (Participants) | 209 | 407
participants with event
  month 4 (122 days) | 10 | 18
  month 8 (244 days) | 22 | 40
  month12 (366 days) | 43 | 74
  month 18 (549 days) | 74 | 117
  month 24 (732 days) | 88 | 145
  month 30 (915 days) | 94 | 156
  month 36 (1098 days) | 94 | 158
Statistical Analysis 1: Comparison: Placebo vs Bosentan; Test type: Superiority or Other; p = 0.2110, Log Rank; Hazard Ratio (HR) = 0.850, 95% CI 2-sided [0.658 to 1.097]

2. Secondary Outcome: Percentage of Patients Who Experienced Either Disease Worsening or Death at 1 Year.
Description: as for outcome 1
Time Frame: 12 months
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants with event
Arm/Group | Placebo | Bosentan
Number analyzed (Participants) | 209 | 407
percentage of participants with event | 23.9 [18.3 to 30.3] | 19.9 [16.1 to 24.1]
Statistical Analysis 1: Comparison: Placebo vs Bosentan; Test type: Superiority or Other; p = 0.2542, Fisher Exact; Relative risk reduction = 0.17, 95% CI 2-sided [-0.13 to 0.39]

ADVERSE EVENTS:
Time Frame: All treatment-emergent adverse events occurring after the start of study treatment and within 24 hours after the end of study treatment
Description: One subject who did not receive study treatment (bosentan) was excluded from the safety population. Events listed as idiopathic pulmonary fibrosis were reported as worsening of idiopathic pulmonary fibrosis.
Arm/Group | Placebo | Bosentan
Serious Adverse Events (participants affected / at risk) | 74/209 | 129/406
Other Adverse Events (participants affected / at risk) | 200/209 | 386/406
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=209) | Bosentan (N=406)
IDIOPATHIC PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 17 | 41
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 6
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 | 4
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 4
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 2
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 0 | 2
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 1
ACUTE INTERSTITIAL PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 0 | 1
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 | 1
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 2 | 0
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PNEUMONIA (Infections and infestations) | 10 | 16
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 5 | 7
BRONCHITIS (Infections and infestations) | 3 | 2
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 1 | 2
APPENDICITIS (Infections and infestations) | 2 | 1
DEVICE RELATED INFECTION (Infections and infestations) | 0 | 1
DIVERTICULITIS (Infections and infestations) | 0 | 1
HERPES ZOSTER OPHTHALMIC (Infections and infestations) | 0 | 1
PILONIDAL CYST (Infections and infestations) | 0 | 1
PYELONEPHRITIS (Infections and infestations) | 0 | 1
UROSEPSIS (Infections and infestations) | 0 | 1
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 | 0
LOBAR PNEUMONIA (Infections and infestations) | 2 | 0
ANAL ABSCESS (Infections and infestations) | 1 | 0
ARTHRITIS BACTERIAL (Infections and infestations) | 1 | 0
CELLULITIS (Infections and infestations) | 1 | 0
HERPES ZOSTER OTICUS (Infections and infestations) | 1 | 0
TRACHEOBRONCHITIS (Infections and infestations) | 1 | 0
URINARY TRACT INFECTION (Infections and infestations) | 1 | 0
VIRAL LABYRINTHITIS (Infections and infestations) | 1 | 0
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 | 6
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 4
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 3
ANGINA UNSTABLE (Cardiac disorders) | 0 | 2
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 3 | 1
CORONARY ARTERY STENOSIS (Cardiac disorders) | 1 | 1
ACUTE CORONARY SYNDROME (Cardiac disorders) | 0 | 1
ATRIAL FLUTTER (Cardiac disorders) | 0 | 1
CARDIAC ARREST (Cardiac disorders) | 0 | 1
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 | 1
ANGINA PECTORIS (Cardiac disorders) | 4 | 0
CARDIAC FAILURE (Cardiac disorders) | 1 | 0
VENTRICULAR HYPOKINESIA (Cardiac disorders) | 1 | 0
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4
BLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
LUNG NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
NON-HODGKIN'S LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 0 | 2
FALL (Injury, poisoning and procedural complications) | 1 | 1
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
EXCORIATION (Injury, poisoning and procedural complications) | 0 | 1
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
RIB FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
TENDON RUPTURE (Injury, poisoning and procedural complications) | 0 | 1
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
CONTUSION (Injury, poisoning and procedural complications) | 1 | 0
HIP FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3 | 3
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 2
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 0 | 1
SJOGREN'S SYNDROME (Musculoskeletal and connective tissue disorders) | 0 | 1
BURSITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
COSTOCHONDRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
FRACTURE NONUNION (Musculoskeletal and connective tissue disorders) | 1 | 0
JOINT EFFUSION (Musculoskeletal and connective tissue disorders) | 1 | 0
POLYARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
SPINAL COLUMN STENOSIS (Musculoskeletal and connective tissue disorders) | 1 | 0
CHEST PAIN (General disorders) | 2 | 2
PYREXIA (General disorders) | 1 | 2
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 | 1
IMPAIRED HEALING (General disorders) | 0 | 1
CHEST DISCOMFORT (General disorders) | 1 | 0
INFLUENZA LIKE ILLNESS (General disorders) | 1 | 0
LIVER FUNCTION TEST ABNORMAL (Investigations) | 0 | 4
PULMONARY FUNCTION TEST DECREASED (Investigations) | 0 | 2
COLITIS (Gastrointestinal disorders) | 0 | 1
COLONIC POLYP (Gastrointestinal disorders) | 0 | 1
GASTRITIS (Gastrointestinal disorders) | 0 | 1
VOMITING (Gastrointestinal disorders) | 0 | 1
ANAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
DIVERTICULUM INTESTINAL HAEMORRHAGIC (Gastrointestinal disorders) | 1 | 0
DYSKINESIA OESOPHAGEAL (Gastrointestinal disorders) | 1 | 0
INGUINAL HERNIA (Gastrointestinal disorders) | 1 | 0
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 0
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
MESENTERIC ARTERIOSCLEROSIS (Gastrointestinal disorders) | 1 | 0
PERITONITIS (Gastrointestinal disorders) | 1 | 0
SYNCOPE (Nervous system disorders) | 2 | 1
DIZZINESS (Nervous system disorders) | 1 | 1
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 0 | 1
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 | 1
CAROTID ARTERY OCCLUSION (Nervous system disorders) | 1 | 0
DEMENTIA (Nervous system disorders) | 1 | 0
HAEMORRHAGIC STROKE (Nervous system disorders) | 1 | 0
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1 | 0
SOMNOLENCE (Nervous system disorders) | 1 | 0
HAEMATURIA (Renal and urinary disorders) | 0 | 3
RENAL MASS (Renal and urinary disorders) | 0 | 1
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 | 2
HYPOTENSION (Vascular disorders) | 1 | 1
INTERMITTENT CLAUDICATION (Vascular disorders) | 0 | 1
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 0 | 1
HYPERTENSION (Vascular disorders) | 1 | 0
TEMPORAL ARTERITIS (Vascular disorders) | 1 | 0
VASCULITIS (Vascular disorders) | 1 | 0
ANAEMIA (Blood and lymphatic system disorders) | 0 | 1
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 | 1
MENIERE'S DISEASE (Ear and labyrinth disorders) | 0 | 1
VERTIGO (Ear and labyrinth disorders) | 0 | 1
BILE DUCT STONE (Hepatobiliary disorders) | 0 | 1
CHOLELITHIASIS (Hepatobiliary disorders) | 0 | 1
HEPATITIS ACUTE (Hepatobiliary disorders) | 0 | 1
CHOLECYSTITIS (Hepatobiliary disorders) | 2 | 0
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 1 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 1
HYPOVOLAEMIA (Metabolism and nutrition disorders) | 0 | 1
CHOLECYSTECTOMY (Surgical and medical procedures) | 0 | 1
TRANSURETHRAL PROSTATECTOMY (Surgical and medical procedures) | 0 | 1
LUNG TRANSPLANT (Surgical and medical procedures) | 1 | 0
ALLERGIC OEDEMA (Immune system disorders) | 0 | 1
DRUG HYPERSENSITIVITY (Immune system disorders) | 0 | 1
ANXIETY (Psychiatric disorders) | 0 | 1
DEPRESSION (Psychiatric disorders) | 0 | 1
PANIC DISORDER (Psychiatric disorders) | 0 | 1
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 0 | 1
PROSTATISM (Reproductive system and breast disorders) | 1 | 0
PRURITUS ALLERGIC (Skin and subcutaneous tissue disorders) | 0 | 1
GOITRE (Endocrine disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=209) | Bosentan (N=406)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 59 | 114
IDIOPATHIC PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 59 | 92
COUGH (Respiratory, thoracic and mediastinal disorders) | 51 | 78
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 24 | 57
FATIGUE (General disorders) | 15 | 46
BRONCHITIS (Infections and infestations) | 28 | 44
HEADACHE (Nervous system disorders) | 22 | 44
NASOPHARYNGITIS (Infections and infestations) | 22 | 40
SINUSITIS (Infections and infestations) | 18 | 38
OEDEMA PERIPHERAL (General disorders) | 23 | 37
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 17 | 30
NAUSEA (Gastrointestinal disorders) | 15 | 27
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 7 | 27
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 18 | 26
LIVER FUNCTION TEST ABNORMAL (Investigations) | 0 | 26
DIZZINESS (Nervous system disorders) | 17 | 24
BACK PAIN (Musculoskeletal and connective tissue disorders) | 16 | 24
CHEST PAIN (General disorders) | 12 | 24
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 6 | 23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Actelion, with steering committee, shall complete the review and provide any modifications required to protect Actelion's patent rights and confidential information within sixty (60) days of receipt of the proposed publication. During this period, Investigator shall not permit publication. If Actelion reasonably anticipates filing a patent application claiming an invention arising out of the Study, such publication shall be delayed until after the application is filed.